CLINICAL TRIAL: NCT03602196
Title: In Vivo Assessment of the Elastic Properties of Women's Pelvic Floor During Pregnancy
Acronym: ELASTOPELV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ELASTOPELV
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pregnant women (Experimental): pregnant women with one visit per trimester of pregnancy (14-18 weeks, 24-28 weeks and 34-38 weeks)
  For the ancillary study: non-pregnant nulliparous women
  Interventions: Other: Perineal ultrasound assessment; Other: Peripheral muscles assessment; Other: Clinical pelvic floor assessment

INTERVENTIONS:
Other: Perineal ultrasound assessment — women were assessed in lithotomy position with an empty bladder at rest, perineal contraction and Valsalva maneuver using a linear translabial probe. We measure the distance between symphysis and ano-rectal angle. In the same position we investigate the levator ani viscoelastic properties using shear wave elastography at rest, Valsalva maneuver and maximal contraction. During the same examination, we assess the viscoelastic properties of the external anal sphincter using shear wave elastography for the 3 conditions: rest, Valsalva, contraction.
  This pelvic floor muscles assessment is performed for each of the three planned visits
  For the ancillary study on non pregnant women: viscoelastic properties of levator ani are assessed at rest, stretch and contraction using shear wave elastography.
  This pelvic floor muscle assessment is performed for each of the two planned visit in the ancillary study.
Other: Peripheral muscles assessment — The visco elastic properties of the biceps brachii muscle and the gastrocnemius medialis muscle are assessed rest, stretch and maximal contraction using shear wave elastography.
  This peripheral muscle assessment is perform for each of the three planned visits.
  For the ancillary study on non pregnant women: viscoelastic properties of biceps brachii and gastrocnemius medialis muscles are assessed at rest, stretch and contraction using shear wave elastography.
  This peripheral muscles ultrasound assessment is performed for each of the two planned visit in the ancillary study.
Other: Clinical pelvic floor assessment — Women undergo a pelvic floor assessment using the Pelvic organ prolapse quantification system. Such an assessment is performed for each of the three planned visits.
  Women included in the ancillary study are not involved with this examination

SUMMARY:
The investigators hypothesize that optimize our risk prediction for pelvic floor disorders after childbirth by taking into account intrinsic women's pelvic floor characteristics and their changes during pregnancy. Shear Wave Elastography (SWE) is a new technology that allowed an in vivo assessment of elastic properties of tissues. The main endpoint of this study is to describe biomechanical changes that occurs into women's pelvic floor during pregnancy using SWE technology.

An ancillary study will investigate the reproducibility of the assessement of the viscoelastic properties of the levator ani muscle, the biceps brachii muscle and the gastrocnemius medialis muscle using shear wave elastography in a nulliparous non-pregnant women cohort

DETAILED DESCRIPTION:
Each woman included in the princeps study undergo 3 visits during pregnancy (14-18 weeks, 24-28 weeks and 34-38 weeks).

Each visit contain a clinical pelvic floor assessment (POP-Q), an ultrasound pelvic floor assessment, an ultrasound pelvic floor muscles (levator ani and external anal sphincter) viscoelastic properties assessment using shear wave elastography and an ultrasound peripheral muscles (biceps brachii and gastrocnemius medialis) using shear wave elastography.

The main objective is to describe changes in viscoelastic properties of pelvic floor muscles during pregnancy. Secondary objectives are to compare muscular behavior of pelvic floor muscles and peripheral muscles during pregnancy.

Data about the delivery are also collected in order to analyse preliminary data about the hypothetic association between viscoelastic properties of women's pelvic floor and both mode of delivery and perineal trauma at childbirth.

An ancillary study involve non-pregnant nulliparous women in oder the investigate the reproducibility of shear wave elastography assessment of the levator ani muscle. Secondary objective is to investigate this reproducibility for biceps brachii and gastrocnemius medialis muscles.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous pregnant women
* Age >18 years
* Normal pregnancy
* BMI < 35 Kg.m-2
* Without previous pelvic floor disorders
* Without muscular diseases, psychiatric diseases

Exclusion Criteria:

* Parous women
* Previous pelvic floor disorders
* BMI > 35 Kg.m-2
* Age < 18 years
* Psychiatric diseases, muscular diseases
* Pathological pregnancy

For the ancillary study about the reproducibility on non-pregnant women

Inclusion Criteria:

* Non pregnant women
* Age >18 years
* BMI < 35 Kg.m-2
* Without previous pelvic floor disorders
* Without muscular diseases, psychiatric diseases

Exclusion Criteria:

* Parous women
* Previous pelvic floor disorders
* BMI > 35 Kg.m-2
* Age < 18 years
* Psychiatric diseases, muscular diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-10-02 (Estimated)

PRIMARY OUTCOMES:
Quantify elastic properties of pregnant women pelvic floor muscles and their changes during pregnancy | 14-18 weeks
  Shear wave modulus value measured for each muscles across the pregnancy.
Quantify elastic properties of pregnant women pelvic floor muscles and their changes during pregnancy | 24-28 weeks
  Shear wave modulus value measured for each muscles across the pregnancy.
Quantify elastic properties of pregnant women pelvic floor muscles and their changes during pregnancy | 34-38 weeks
  Shear wave modulus value measured for each muscles across the pregnancy.

SECONDARY OUTCOMES:
Look for an association between shear modulus assessed for pelvic floor muscles and perineal distension assessed by clinical and ultrasound assessment | 14-18 weeks
  Association between the shear modulus assessed for pelvic floor muscles and both clinical (POP-Q) and ultrasound pelvic floor distension.
Look for an association between shear modulus assessed for pelvic floor muscles and perineal distension assessed by clinical and ultrasound assessment | 24-28 weeks
  Association between the shear modulus assessed for pelvic floor muscles and both clinical (POP-Q) and ultrasound pelvic floor distension.
Look for an association between shear modulus assessed for pelvic floor muscles and perineal distension assessed by clinical and ultrasound assessment | 34-38 weeks
  Association between the shear modulus assessed for pelvic floor muscles and both clinical (POP-Q) and ultrasound pelvic floor distension.
Look for an association between changes in elastic properties of pelvic floor muscles and peripheral muscles (biceps brachii and gastrocnemius medialis). | 14-18 weeks
  Association between shear modulus changes assessed for pelvic floor muscles (levator ani and/or external anal sphincter) and shear modulus changes assessed for peripheral muscles (biceps brachii or gastrocnemius medialis)
Look for an association between changes in elastic properties of pelvic floor muscles and peripheral muscles (biceps brachii and gastrocnemius medialis). | 24-28 weeks
  Association between the shear modulus changes assessed for pelvic floor muscles (levator ani and/or external anal sphincter) and shear modulus changes assessed for peripheral muscles (biceps brachii or gastrocnemius medialis)
Look for an association between changes in elastic properties of pelvic floor muscles and peripheral muscles (biceps brachii and gastrocnemius medialis). | 34-38 weeks
  Association between the shear modulus changes assessed for pelvic floor muscles (levator ani and/or external anal sphincter) and shear modulus changes assessed for peripheral muscles (biceps brachii or gastrocnemius medialis)
To assess the feasibility of measuring the viscoelastic properties of the external anal sphincter using shear wave elastography | 14-18 then 24-28 then 34-38 weeks
  Number of success procedures for each visit and each condition
Quantify elastic properties of pregnant women external anal sphincter and their changes during pregnancy | 14-18 then 24-28 then 34-38 weeks
  shear modulus of the external anal sphincter
Investigate if pelvic floor muscle's shear modulus (viscoelastic properties) and their changes during pregnancy are associated with both : the mode of delivery (spontaneous, instrumental, cesarean) and perineal tears occurrence. | Shear modulus measurements (14-18 then 24-28 then 34-38 weeks) and the delivery
  Association between the mode of delivery (spontaneous, instrumental or cesarean), the perineal trauma (perineal tears occurrence) and the shear modulus of pelvic floor muscles and their changes during pregnancy

OTHER OUTCOMES:
Reproducibility of the technique in non pregnant women cohort | 2 examinations spaced from 12 hours at least and 7 days maximally
  Assessment of the intraclass coefficient of correlation and the coefficient of variation for each measurement (levator ani, gastrocnemius medialis, biceps brachii) using shear wave elastography. The comparison is proceed between two examination spaced from at least 12hours and maximal 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand GACHON, Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gachon B, Fritel X, Pierre F, Nordez A. In vivo assessment of the elastic properties of women's pelvic floor during pregnancy using shear wave elastography: design and protocol of the ELASTOPELV study. BMC Musculoskelet Disord. 2020 May 15;21(1):305. doi: 10.1186/s12891-020-03333-y. PMID 32414362